CLINICAL TRIAL: NCT06820944
Title: Theobromine Consumption From Cocoa and Cardiovascular Risk Factors in Humans: Evidence for Health Claims
Brief Title: Theobromine From Cocoa and Cardiovascular Risk Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Siraphat Taesuwan, Assistant Professor, Chiang Mai University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21/67
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: cocoa consumption; theobromine; trimethylamine-n-oxide; crossover; randomized trial; chocolate consumption
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dark chocolate (Experimental): 100 g/day of dark chocolate
  Interventions: Other: dark chocolate
- White chocolate (Placebo Comparator): 80 g/day of white chocolate
  Interventions: Other: white chocolate

INTERVENTIONS:
Other: dark chocolate — Consumption of 100 g/day of 72% dark chocolate bar for 14 days consecutively
  Arms: Dark chocolate
Other: white chocolate — Consumption of 80 g/day of white chocolate bar for 14 days consecutively
  Arms: White chocolate

SUMMARY:
The goal of this clinical trial is to examine whether consumption of dark chocolate affects blood pressure and a cardiovascular risk factor called trimethylamine N-oxide in Thai male participants with hypertension. The main questions it aims to answer are:

Can consumption of dark chocolate lower blood pressure? Can consumption of dark chocolate lower blood trimethylamine N-oxide?

Researchers will compare dark chocolate to white chocolate to see if the effects are due to theobromine (a key bioactive compound in dark chocolate).

Participants will consume either 100 g 72% dark chocolate bar or 80 g white chocolate bar daily for 14 days, rest for 7 days, and then switch to the other type of chocolate.

DETAILED DESCRIPTION:
This is a randomized cross-over trial conducted in Chiang Mai, Thailand. The goal of this clinical trial is to examine whether consumption of dark chocolate affects cardiovascular risk factors, with the primary outcomes being blood pressure and a cardiovascular risk factor called trimethylamine N-oxide. Participants are Thai males aged 35-70 years with hypertension who live in the Chiang Mai area.

42 Participants will consume either 100 g 72% dark chocolate bar (~2.5 servings, providing ~900 mg theobromine) or 80 g white chocolate bar (~2 servings, providing 0 mg theobromine) daily for 14 days. After a 7-day wash-out period, the participant will repeat the protocol with the other intervention.

ELIGIBILITY:
Inclusion criteria

* Male
* Age between 35 to 70 years
* BMI less than 30 kg/m^2
* Systolic blood pressure between 130 to 159 mmHg or Diastolic blood pressure between 85 to 99 mmHg.
* Do not smoke.

Exclusion criteria

* Cannot drink beverages and consume foods that have caffeine.
* Take medicine to lower cholesterol and triglyceride levels, treat high blood pressure, or diabetes.
* Have liver and kidney inflammation.
* Use antibiotics within 1 month of study.
* Use choline or probiotic supplements regularly within 1 month of study.
* Consume more than 30 alcoholic drinks per week.
* Have chronic diseases.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender males and transgender males who do not take female hormones
Enrollment: 42 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Measured at the beginning and the end of each intervention period (14 days)
  Office blood pressure measured in the morning after fasting
Fasting blood trimethylamine-N-oxide | Measured at the beginning and the end of each intervention period (14 days)
  Fasting blood trimethylamine-n-oxide concentrations

SECONDARY OUTCOMES:
Postprandial trimethylamine-N-oxide | Measured at the beginning and the end of the dark chocolate intervention (14 days)
  Urinary trimethylamine-N-oxide concentrations at 24 and 48 hours after consumption of a test meal (3 boiled eggs)
Ankle-brachial index | From the beginning and end of each intervention period of 14 days
  Ankle-brachial index is a noninvasive test that measures the ratio of blood pressure in the ankle to the blood pressure in the arm.

CONTACTS AND LOCATIONS:
Overall Officials: Kongsak Boonyapranai, Doctoral degree, Principal Investigator — Research Institute for Health Science, Chiang Mai University
Locations (1):
- Research Institute for Health Sciences, Chiang Mai University, Mueang, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Chocolate consumption and cardiometabolic disorders: systematic review and meta-analysis. BMJ, 343(7825). — https://doi.org/10.1136/BMJ.D4488
- See also: The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Research, 28(2), 193-213. — https://doi.org/10.1016/0165-1781(89)90047-4
- See also: Effect of dark chocolate on flow-mediated dilatation: Systematic review, meta-analysis, and dose-response analysis of randomized controlled trials. Clinical Nutrition ESPEN, 36, 17-27. — https://doi.org/10.1016/J.CLNESP.2019.10.017
- See also: Effects of chocolate, cocoa, and flavan-3-ols on cardiovascular health: a systematic review and meta-analysis of randomized trials. The American Journal of Clinical Nutrition, 95(3), 740-751. — https://doi.org/10.3945/AJCN.111.023457
- See also: Impact of cocoa flavanols on human health. Food and Chemical Toxicology, 151, 112121. — https://doi.org/10.1016/J.FCT.2021.112121
- See also: Effect of cocoa and theobromine consumption on serum HDL-cholesterol concentrations: A randomized controlled trial. American Journal of Clinical Nutrition, 97(6), 1201-1209. — https://doi.org/10.3945/ajcn.112.047373
- See also: (2016). Relationship of Serum Trimethylamine N-Oxide (TMAO) Levels with early Atherosclerosis in Humans. Scientific Reports, 6(1), 26745. — https://doi.org/10.1038/srep26745
- See also: (2019). Chocolate consumption and risk of cardiovascular diseases: a meta-analysis of prospective studies. Heart, 105(1), 49-55. — https://doi.org/10.1136/HEARTJNL-2018-313131
- See also: Dose-response relationship between cocoa flavanols and human endothelial function: a systematic review and meta-analysis of randomized trials. Food & Function, 10(10), 6322-6330. — https://doi.org/10.1039/C9FO01747J
- See also: ). Effects of cocoa products/dark chocolate on serum lipids: a meta-analysis. European Journal of Clinical Nutrition 2011 65:8, 65(8), 879-886. — https://doi.org/10.1038/ejcn.2011.64